CLINICAL TRIAL: NCT04367324
Title: Effect of Low-Level Laser Therapy Following Direct Pulp Capping on Postoperative Sensitivity by Thermal Stimulus: A Retrospective Study
Brief Title: Effect of Low-Level Laser Therapy Following Direct Pulp Capping on Postoperative Sensitivity by Thermal Stimulus
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Adem Günaydin, Research Assistant, Ordu University
Other Study IDs: Ordu
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Low-level Laser Therapy
Keywords: direct pulp capping; low level laser therapy; thermal stimulus; biostimulation
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low level laser therapy: Applied the low-level laser irradiation
  Interventions: Device: Low-level laser therapy
- Control: No low-level laser application

INTERVENTIONS:
Device: Low-level laser therapy — The low-level laser was applied to each patient in low-level laser therapy group.
  Groups: Low level laser therapy

SUMMARY:
The aim of this study was to investigate the effect of low-level laser therapy (LLLT) on postoperative pain provoked by thermal stimulation in direct pulp capping. All the patients who received consent form in this retrospective study were retrieved from the records of patients attended for routine dental treatment at the Ordu University, Faculty of Dentistry, Department of Endodontics between 01.10.2017-01.10.2018. Study subjects were recruited from the pool of patients who performed direct pulp capping by a single operator. A total of 123 pre-treated teeth of 123 patients who referred to Ordu University, Faculty of Dentistry were examined. Follow-up examinations were carried out at postoperative 6th hours, 1st and 7th days with visual analog scale (VAS), and treatment outcome were assessed. Participants were allocated to the laser and control group which consist of 42 patients in each group. 6 patients were excluded from the study due to missing data in both groups. Thus, data from 72 patients who had been carried out direct pulp capping were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Mandibular and maxillary permanent molars with pulpal exposure between 0.5-1.0 mm
2. Periodontally healthy teeth (no more than 3mm probing depth)
3. Pulpal exposure occurring only on the occlusal side of the tooth
4. Systemically healthy participant
5. Participants who signed the written consent form
6. Patients aged 15-45
7. Patients who have not used analgesic or antibiotic in the past two weeks
8. Patients whose data are fully and accurately recorded
9. Patients who do not use immunosuppressive drugs and do not need antibiotic prophylaxis

Exclusion Criteria:

1. Patients who need a second anesthetic
2. Presence of a previous restoration of the tooth
3. Patients using psychiatric or sedative medication
4. Patients who had a direct pulp capping treatment on several teeth
5. Patients with tooth pain and unable to localize this pain
6. Patients taking pain medication within 1 week after the procedures
7. Patients with a lack of data during follow-up
8. Treated teeth without following clinical procedures

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All the participants in this study were retrieved from the pool of patients who attended for routine treatment at the Department of Endodontics at the University Hospital of Ordu between October 2017 and October 2018. Those patients who had received DPC treatment by a single operator were selected.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Effect of low-level laser therapy following direct pulp capping on postoperative sensitivity as assessed by visual analog scale. | 7 days
  Postoperative sensitivity was assessed and documented via a visual analog scale. The visual analog scale consists of a 100 mm line which is represented at one end by a sign 'no pain' and at the other end 'unbearable pain'. This form was given to each patient and instructed to mark at home according to the pain intensity at 6th hours. Also, patients were seen 1 and 7 days postoperatively to mark the degree of pain on the visual analog scale. Patients were informed that the marking must be performed only when sensitivity induced by the cold stimulus. On a visual analog scale named postoperative sensitivity scale, '0' presents the minimum value and '10' presents the maximum value. High scores indicate a worse result, while low scores indicate a better result. Lower sensitivity was detected on the visual analog scale at 7th days in the low-level laser therapy group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Günaydın, Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
undecided